CLINICAL TRIAL: NCT03689543
Title: The Effects of an ER Beta Agonist (Lilly Compound LY500307) on Estradiol-withdrawal-induced Mood Symptoms in Women With Past Perimenopausal Depression
Brief Title: Estrogen Receptor Beta and Mood
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 180144; 18-M-0144
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08-15

CONDITIONS: Perimenopause-Related Depression
Keywords: Perimenopause-related depression
MeSH Terms: interventions — Estradiol; erteberel; Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: High dose LY500307 compound (Experimental): Female participants received open label estradiol 0.1mg transdermal patch per day for three weeks. Then participants received LY500307 compound 75mg orally once per day for three weeks under double blind conditions. Participants with a uterus received Provera 5mg orally once a day for one week after completion of randomization.
  Interventions: Drug: Estradiol; Drug: ER Beta Agonist; Drug: Provera
- Arm 2: Low dose LY500307 compound (Active Comparator): Female participants received open label estradiol 0.1mg transdermal patch per day for three weeks. Then participants received a combination of LY500307 compound 25mg and placebo orally once per day for three weeks under double blind conditions. Participants with a uterus received Provera 5mg orally once a day for one week after completion of randomization.
  Interventions: Drug: Estradiol; Drug: ER Beta Agonist; Other: Placebo; Drug: Provera
- Arm 3: Placebo (Placebo Comparator): Female participants received open label estradiol 0.1mg transdermal patch per day for three weeks. Then participants received placebo orally once per day for three weeks under double blind conditions. Participants with a uterus received Provera 5mg orally once a day for one week after completion of randomization.
  Interventions: Drug: Estradiol; Other: Placebo; Drug: Provera

INTERVENTIONS:
Drug: Estradiol — Estradiol patch 0.1 mg transdermal every three days for three weeks
Drug: ER Beta Agonist — Lilly Compound LY500307, a selective estrogen receptor (ER) beta agonist
  Other Names: LY500307
  Arms: Arm 1: High dose LY500307 compound; Arm 2: Low dose LY500307 compound
Other: Placebo — Placebo orally once daily
  Arms: Arm 2: Low dose LY500307 compound; Arm 3: Placebo
Drug: Provera — Provera 5 mg orally once a day for one week after completion of randomization

SUMMARY:
Background:

Our previous studies have found that women who had depression during the perimenopause may have mood symptoms again if they stop estrogen therapy. Estrogen acts in the brain and other tissues by binding to estrogen receptors. There are two main types of estrogen receptors. They are estrogen receptor alpha and beta. Several studies have shown that estrogen receptor beta may play an important role in anxiety- and depressive-like behaviors in animals.

Objectives:

To examine a possible mechanism mediating the effects of estradiol-withdrawal on mood symptoms in asymptomatic postmenopausal women with a past perimenopausal depression. To evaluate the efficacy and safety of a selective estrogen receptor (ER) beta agonist (Lilly Compound LY500307) to prevent estradiol withdrawal-induced mood symptoms.

Eligibility:

Healthy, non-depressed postmenopausal women, ages 45 to 65, with a well-documented past perimenopause-related depression (within 12 years) and whose mood systems got better with estradiol

Design:

Participants will be screened with:

Medical history

Physical exam

Blood tests

Psychiatric interview

Gynecological exam

* Participants able to get pregnant must use effective barrier birth control throughout the study.
* During the first 3 weeks, participants will wear an estrogen patch. It is 1x2 inches and will be replaced every 3 days.
* For the next 3 weeks, participants will take 3 study capsules every morning. They will not know if they get the study drug or placebo.
* Some participants will also take a progesterone-like drug for 1 week at the end of the medication phase of the study.
* Participants will have 9 one-hour study visits. They will have blood samples and vital signs taken. They will answer questions about mood and behavior symptoms.
* Participants will keep a daily log of these symptoms.
* Participants will have 2 transvaginal ultrasounds. A probe is temporarily placed 2-3 inches into the vaginal canal and sound waves are used to create pictures of the lining of the uterus.
* Participants will have a final visit 4 weeks after stopping the study drug. They will answer questions about mood and side effects.

DETAILED DESCRIPTION:
OBJECTIVE:

Depression risk increases during the perimenopause, and depression is cited as a primary reason for resuming menopausal hormone therapy (HT). Community-based epidemiologic studies document a 1.5-3 fold greater risk of first onset and recurrent depressions in women during the perimenopause compared with those who are premenopausal (or who are several years postmenopausal). Observational studies report the emergence of depressive symptoms after the discontinuation of HT in 5-10% of women. The role of estradiol (E2) - either declining or low levels - in the precipitation of perimenopausal depression (PMD) is unknown, largely due to the associational and indirect nature of the evidence linking ovarian function and depression. In study 03-M-0175, our results demonstrated that estradiol withdrawal was associated with a significant increase in depressive symptoms in those women with a past depression during the perimenopause. Of note, the effects of estradiol primarily occur through activation of two receptor subtypes, often with opposing outcomes: estrogen receptor (ER) alpha, and ER beta. Therefore, in this protocol, we examined the ability of a selective ER beta agonist (LY500307) to prevent estradiol withdrawal- induced mood symptoms in women with past perimenopausal depression. We focused on ER beta because the beta estrogen receptor is reported to mediate the effects of estradiol on the serotonergic system and mediate the antidepressant-like effects of estradiol in the forced-swim test. Moreover, selective agonists of estrogen receptor beta have been demonstrated to attenuate the behavioral and hypothalamic-pituitary-adrenal (HPA) axis response to stress.

Our objective is to examine the specific role of estrogen receptor beta in the effects of estrogen withdrawal in women with a past perimenopause-related depression. Results of this study will determine the role of ER beta in estradiol withdrawal-induced mood symptoms and can provide preliminary data to support the efficacy and safety of this compound as a treatment for depression during the perimenopausal transition.

STUDY POPULATION:

Healthy, non-depressed postmenopausal women, ages 45 to 65, with a well-documented past perimenopause-related depression (within 12 years) and whose mood systems got better with estradiol

DESIGN:

The medication phase of this study is a seven-week randomized, double blind, placebo controlled study and there is a four week follow-up evaluation phase to monitor all women for the emergence of adverse effects post-medication exposure. Participants will have weekly outpatient visits, weekly blood draws and will also complete daily symptom rating scales. The study involves a three week baseline phase in which all women receive open label (OL) estradiol therapy (ET) at a dose of 100 micrograms per day by transdermal skin patch, after which all women receive three weeks of double blind (DB) medication (i.e., LY500307 [at a daily dose of either 25 mg or 75 mg] or placebo). All participants will receive three capsules of LY500307 or placebo each morning consisting of the following formulations: 1) women randomized to 75 mg LY500307 will receive three capsules each containing 25 mg LY500307; 2) women randomized to 25 mg LY500307 will receive one capsule containing 25 mg LY500307 and two capsules of placebo; and 3) women randomized to placebo will receive three capsules each containing placebo. Then, in non-menstruating women (i.e., the absence of reported menstrual bleeding of greater than 1-2 days during the double blind phase of this study), the double blind phase will be followed by one week of Provera to precipitate a progestin-induced menses. The week of Provera is not a research-related intervention but is clinically-indicated to induce endometrial shedding that will eliminate potentially abnormal endometrial tissue consequent to the three weeks of unopposed estradiol exposure.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Women with a past perimenopause-related depression (within 12 years). The diagnosis of perimenopause-related depression will be based on a history of a past depressive episode (major or minor depression confirmed by Structured Clinical Interview for Diagnostic and Statistical Manual (DSM)-V (SCID)) at midlife in association with menstrual cycle irregularity (and possibly hot flushes and/or vaginal dryness) and in whom menopausal hormone therapy was reported to improve their depression at any time within the prior twelve years. All women participating in this protocol will be screened with psychiatric, medical, and reproductive evaluations to confirm they are in good medical health.
2. Age 45 to 65
3. Medication free (including no mood stabilizers, no sleep medication) except for the following: women on menopausal hormone therapy who will discontinue these medications at the start of this study and have their hormone therapy replaced with estradiol 100mcg per day (as described below), women who are on stable doses of thyroid replacement for at least six months prior to study enrollment, or women who occasionally take non-steroidal anti-inflammatory drugs [NSAIDs] or allergy medications (although we will ask women to minimize the use of these medications during the study).
4. Subjects must have consent capacity

EXCLUSION CRITERIA:

The following conditions will constitute contraindications to participate in this protocol:

1. Any current Axis 1 psychiatric illness or any clinically significant sleep disorder;
2. Women with histories of hormone replacement therapy-induced dysphoria due to either the estrogen or the progesterone components of their hormone replacement;
3. Past history of major depression with suicidal ideation;
4. History of ischemic cardiac disease, pulmonary embolism, or thrombophlebitis;
5. Renal disease; hepatic dysfunction; history of cholecystitis; hypertension;
6. Women with a history of carcinoma of the breast or any undiagnosed breast nodule/mass;
7. Women with a history of uterine cancer, ill-defined pelvic lesions, particularly undiagnosed ovarian enlargement, undiagnosed vaginal bleeding;
8. Pregnant women; sexually active women will be required to employ barrier contraceptive methods;
9. Cerebrovascular disease (stroke);
10. Recurrent migraine headaches;
11. Women who have had a hysterectomy before one year after their last menstrual period.

National Institute of Mental Health (NIMH) employees/staff and their immediate family members will be excluded from the study per NIMH policy.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Schmidt, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with database of Genotypes and Phenotypes (dbGaP), Biomedical Translational Research Information System (BTRIS) and NIMH Data Archive as determined by the Principal Investigator.
Supporting Information: Study Protocol, ICF
Time Frame: Starting 24 months after final publication
Access Criteria: Data will be shared with dbGaP, BTRIS and NIMH Data Archive as determined by the Principal Investigator.

REFERENCES:
- [Background] Cohen LS, Soares CN, Vitonis AF, Otto MW, Harlow BL. Risk for new onset of depression during the menopausal transition: the Harvard study of moods and cycles. Arch Gen Psychiatry. 2006 Apr;63(4):385-90. doi: 10.1001/archpsyc.63.4.385. PMID 16585467
- [Background] Freeman EW, Sammel MD, Lin H, Nelson DB. Associations of hormones and menopausal status with depressed mood in women with no history of depression. Arch Gen Psychiatry. 2006 Apr;63(4):375-82. doi: 10.1001/archpsyc.63.4.375. PMID 16585466
- [Background] Freeman EW. Associations of depression with the transition to menopause. Menopause. 2010 Jul;17(4):823-7. doi: 10.1097/gme.0b013e3181db9f8b. PMID 20531231
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-M-0144.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: of the 74 participants consented to study, 19 participants failed screening and nine (9) dropped out prior to randomization
Period: Overall Study
Arm/Group | Arm 1: High Dose LY500307 Compound | Arm 2: Low Dose LY500307 Compound | Arm 3: Placebo
Started | 15 | 15 | 16
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: High Dose LY500307 Compound | Arm 2: Low Dose LY500307 Compound | Arm 3: Placebo | Total
Number analyzed (Participants) | 15 | 15 | 16 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 16 | 46
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 16 | 46
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 3 | 5
  Not Hispanic or Latino | 15 | 12 | 13 | 40
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 5
  White | 13 | 11 | 12 | 36
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Center for Epidemiologic Studies-Depression (CES-D) Scale Mean Total Score
Description: Center for Epidemiologic Studies-Depression (CES-D) Scale is a 20-item questionnaire that asks participants to rate how often over the past week they experienced symptoms associated with depression. Each item is rated from 0 to 3 (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Total scores range from 0 to 60, with high scores indicating greater depressive symptoms. CES-D scores >8 and <16 is consistent with subsyndromal depression. CES-D scores > 16 are consistent with clinically significant depressive symptoms of at least moderate severity. Participants completed the CES-D at baseline and every week for six weeks during each of the study phases (open label estradiol patch, double blind placebo or LY500307 compound). Analysis was calculated as the mean of scores for baseline (week 0) and weekly through week six (6).
Time Frame: Baseline, then weekly through end of week six
Population: All participants who were randomized to arms in the study. One participant dropped out at week 5 therefore did not complete week 6 questionnaire.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm 1: High Dose LY500307 Compound | Arm 2: Low Dose LY500307 Compound | Arm 3: Placebo
Number analyzed (Participants) | 15 | 15 | 16
Units on a scale
  Baseline | 12.96 (9.06) | 18.02 (11.27) | 11.53 (9.03)
  Week 1 | 9.43 (7.11) | 10.67 (8.01) | 5.38 (6.83)
  Week 2 | 4.27 (4.22) | 5.60 (4.70) | 3.44 (3.83)
  Week 3 | 3.47 (4.09) | 4.13 (3.87) | 2.25 (2.82)
  Week 4 | 5.60 (5.45) | 5.27 (5.08) | 5.19 (7.20)
  Week 5 | 7.47 (11.36) | 5.47 (5.18) | 8.25 (9.55)
  Week 6: number analyzed (Participants) | 15 | 15 | 15
  Week 6 | 8.40 (11.19) | 6.00 (6.37) | 9.93 (9.32)

2. Primary Outcome: Hamilton Rating Scale of Depression (HRSD) Mean Total Score
Description: The Hamilton Rating Scale of Depression (HRSD) is a 21-item scale used by clinicians to assess the severity of depressive symptoms administered through a structured interview. The HRSD contains 21 items, but four questions are not added to the numerical total score. The first 17 items are scored on a 3 (0-2) or 5 (0-4) point scale, with total score range between 0 and 52. Higher score indicates greater depressive symptom. Scores of 0-7 are considered normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression. Participants completed the HRSD at baseline and every week for six weeks during each of the study phases (open label estradiol patch, double blind placebo or LY500307 compound). Analysis was calculated as the mean of scores for baseline (week 0) and weekly through week six (6).
Time Frame: Baseline, then weekly through end of week six
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm 1: High Dose LY500307 Compound | Arm 2: Low Dose LY500307 Compound | Arm 3: Placebo
Number analyzed (Participants) | 15 | 15 | 16
Units on a scale
  Baseline | 5.78 (4.84) | 5.92 (3.45) | 3.59 (2.81)
  Week 1 | 3.87 (4.1) | 2.87 (2.92) | 2.63 (3.07)
  Week 2 | 1.93 (1.94) | 1 (1.31) | 0.69 (0.95)
  Week 3 | 0.87 (1.06) | 0.73 (0.7) | 0.69 (0.79)
  Week 4 | 2.93 (3.28) | 3.07 (3.37) | 2.94 (2.79)
  Week 5 | 4 (7.03) | 3.6 (3.76) | 5.25 (5.52)
  Week 6: number analyzed (Participants) | 15 | 15 | 15
  Week 6 | 5.52 (7.17) | 3.8 (3.67) | 4.87 (4.69)

ADVERSE EVENTS:
Time Frame: 4-5 weeks after completion of interventions, for a maximum of 11 weeks from start of study.
Groups:
- Estradiol Transdermal Patch: Female participants received open label estradiol 0.1mg transdermal patch per day for three weeks.
- Arm 1: High Dose LY500307 Compound: Female participants received LY500307 compound 75mg orally once per day for three weeks under double blind conditions.
- Arm 2: Low Dose LY500307 Compound: Female participants received a combination of LY500307 compound 25mg and placebo orally once per day for three weeks under double blind conditions.
- Arm 3: Placebo: Female participants received placebo orally once per day for three weeks under double blind conditions.
- Provera Oral Tablet: Female participants with a uterus received Provera 5mg orally once a day for one week after completion of randomization.
Arm/Group | Estradiol Transdermal Patch | Arm 1: High Dose LY500307 Compound | Arm 2: Low Dose LY500307 Compound | Arm 3: Placebo | Provera Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/15 | 0/15 | 0/16 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/15 | 0/15 | 0/16 | 0/42
Other Adverse Events (participants affected / at risk) | 6/46 | 3/15 | 2/15 | 1/16 | 3/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Estradiol Transdermal Patch (N=46) | Arm 1: High Dose LY500307 Compound (N=15) | Arm 2: Low Dose LY500307 Compound (N=15) | Arm 3: Placebo (N=16) | Provera Oral Tablet (N=42)
Cardiac flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diverticulitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Oestradiol increased (Investigations) | 0 | 0 | 1 | 0 | 0
SARS-CoV-2 test (Investigations) | 1 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Uterine disorder (Reproductive system and breast disorders) | 3 | 0 | 0 | 0 | 0
Nodular rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03689543/Prot_SAP_000.pdf